CLINICAL TRIAL: NCT04748198
Title: Effect of Intracorneal Ring Segments on Posterior Corneal Tomography in Eyes With Keratoconus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMASU MD 140/2018
Record Dates: First submitted 2021-01-31; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Keratoconus; Keratoconus Posterior
Keywords: keratoconus; intracorneal ring segments; posterior corneal surface
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Intracorneal ring segments are implanted for treatment of keratoconus, and posterior corneal surface is assessed preoperatively and postoperatively.
  Interventions: Procedure: Intracorneal ring segment implantation

INTERVENTIONS:
Procedure: Intracorneal ring segment implantation — Surgical procedure for keratoconus treatment. A tunnel is created in the corneal stroma with femtosecond laser and ring segments are implanted in the corneal stroma

SUMMARY:
Our purpose is to analyze the changes induced in the posterior corneal surface in patients implanted with intracorneal ring segments for treatment of keratoconus. Patients are assessed with corneal imaging device preoperatively and at 1, 3, 6 and 12 months postoperatively.

DETAILED DESCRIPTION:
Procedure: Femtosecond laser assisted implantation of intracorneal ring segments in keratoconus patients Uncorrected visual acuity (UCVA), best corrected visual acuity (BCVA), refraction, keratometric (K) readings of the anterior and posterior surface, corneal asphericity (Q value) of the anterior and posterior surface, and anterior and posterior elevations are evaluated using a corneal imaging device preoperatively and at 1, 3, 6 and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria

* Patients with keratoconus grade 1, 2 or 3 according to Amsler-Krumeich classification.
* Best corrected visual acuity (BCVA) ≤ 6/12.
* Mean front keratometric (K) readings ≤ 60 diopters (D).
* Corneal thickness ≥ 400 µm at the location of ICRS implantation.
* Clear central cornea

Exclusion Criteria

* Central corneal opacity.
* Previous corneal laser refractive surgery.
* Previous corneal collagen cross linking.
* Previous cataract surgery or phakic IOL implantation.
* History of herpetic keratitis.
* History of acute hydrops.
* Ocular comorbidities such as cataract, glaucoma or retinal disease.
* Systemic diseases affecting healing process such as autoimmune or connective tissue disease.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Posterior corneal astigmatism | Baseline to 12 months
  It is measured by corneal imaging device preoperatively and postoperatively

SECONDARY OUTCOMES:
Visual Acuity | Baseline to 12 months
  It is measured by Snellen Chart Acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sogutlu E, Pinero DP, Kubaloglu A, Alio JL, Cinar Y. Elevation changes of central posterior corneal surface after intracorneal ring segment implantation in keratoconus. Cornea. 2012 Apr;31(4):387-95. doi: 10.1097/ICO.0b013e31822481df. PMID 22410615
- [Background] Muftuoglu O, Aydin R, Kilic Muftuoglu I. Persistence of the Cone on the Posterior Corneal Surface Affecting Corneal Aberration Changes After Intracorneal Ring Segment Implantation in Patients With Keratoconus. Cornea. 2018 Mar;37(3):347-353. doi: 10.1097/ICO.0000000000001492. PMID 29256982
- [Background] Rho CR, Na KS, Yoo YS, Pandey C, Park CW, Joo CK. Changes in anterior and posterior corneal parameters in patients with keratoconus after intrastromal corneal-ring segment implantation. Curr Eye Res. 2013 Aug;38(8):843-50. doi: 10.3109/02713683.2013.788723. Epub 2013 Apr 22. PMID 23806046

DOCUMENTS (1):
  • Study Protocol (2018-05-30): https://cdn.clinicaltrials.gov/large-docs/98/NCT04748198/Prot_000.pdf